CLINICAL TRIAL: NCT02407912
Title: Intrapleural Hypertonic Cisplatin Treatment for Malignant Pleural Effusion in Patients With Non-small-cell Lung Cancer.
Brief Title: Cisplatin for Malignant Pleural Effusion in Patients With Non-small-cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Hongbiao Wang, Associate chief physician, Shantou University Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LXY 01
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin (Experimental): 75 mg of body surface area of ciplatin in distilled water is injected in to the chest through a chesttube.
  Interventions: Drug: cisplatin
- Control (No Intervention): No intervention was applied.

INTERVENTIONS:
Drug: cisplatin — ciplatin in distilled water is injected into the chest for 48 h.
  Other Names: cisplatinum
  Arms: Cisplatin

SUMMARY:
To assess the effect and toxicity of intrapleural administration of hypertonic cisplatin for malignant pleural effusion in patients with non-small-cell lung cancer.

DETAILED DESCRIPTION:
The lung was fully expanded by a thoracostomy using a chest tube with a double lumen, and then the patients were enrolled into the trial.First, premedication including antiemetics and hydration were performed. Thereafter, 75 mg of body surface area of cisplatin in 50 ml of distilled water was injected through a chest tube.The patients were asked to change position (supine and bilateral decubital) from time to time for 30 minutes. The chest tube was clamped for 48 h and then the tube was declamped and allowed to drain. When the drainage effusion was less than 100 ml a day, the chest tube was removed. Any patient whose drainage effusion continued for over 2 weeks was withdrawn from the trial and was also judged to be a nonresponder.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically proven and previously untreated malignant pleural effusion of Non-small-cell Lung Cancer;
* An Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1;
* A leucocyte count of≥4000µl;
* A platelet count of≥100000µl;
* A normal creatinine level;
* Serum glutamic oxaloacetic transaminase/glutamic pyruvic transaminase levels of no more than twice the upper limit of normal;
* Survival time ≥12 weeks.

Exclusion Criteria:

* Previously treated malignant pleural effusion;
* Pericardial effusion；
* Pregnant；
* Uncontrolled hypertension or diabetes；
* Liver cihrosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
overall response rate | one month

CONTACTS AND LOCATIONS:
Overall Officials: Hongbiao Wang, Master, Principal Investigator — Affiliated Cancer Hospital of Shantou University Medical College
Locations (1):
- Department of medical oncology, Shantou, Guangdong, China